CLINICAL TRIAL: NCT00099996
Title: A Study to Assess Adding Ezetimibe 30 mg to Ongoing Treatment With Ezetimibe 10 mg in Patients With Homozygous Sitosterolemia
Brief Title: Higher-Dose Ezetimibe to Treat Homozygous Sitosterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050060; 05-H-0060
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-12

CONDITIONS: Heart Diseases; Metabolism, Inborn Errors
Keywords: Sitosterolemia; Sitosterol; Ezetimibe; Absorption; Intestine; Cholesterol; Atherosclerosis; Homozygous Sitosterolemia
MeSH Terms: conditions — Heart Diseases; Metabolism, Inborn Errors; Sitosterolemia; Atherosclerosis | interventions — Ezetimibe

INTERVENTIONS:
Drug: SCH-58235
Drug: Ezetimibe

SUMMARY:
This study will test the safety and effectiveness of 40 mg of ezetimibe (Zetia ) daily in lowering blood levels of cholesterol and of the plant sterols sitosterol and campesterol in patients with homozygous sitosterolemia, an inherited disorder of sterol metabolism. (Sterols are alcohol substances found in animal and plant fats.) In this disorder, an excess of many plant sterols is absorbed and not enough excreted. Patients can develop atherosclerosis and coronary heart disease as early as childhood, as well as other problems including arthritis, arthralgia, and tendon xanthomas (lipid deposits). Current treatment consists of ezetimibe 10 mg, dietary restriction of plant and shellfish sterols, and bile salt binding resins. Ezetimibe is a cholesterol-lowering drug that inhibits intestinal absorption of cholesterol and structurally related plant sterols across the intestinal wall.

Patients with homozygous sitosterolemia who are between 18 and 85 years of age have completed NHLBI's 1-year study of ezetimibe at 10 mg a day may be eligible for this study.

All participants maintain their current stable diet and take a 10-mg pill of ezetimibe daily for 26 weeks. They are also randomly selected to take either an additional 30-mg pill of ezetimibe or a placebo (look-alike pill with no active ingredients). Patients fast for at least 12 hours before each of 6 visits scheduled during the course of the study. At these visits, patients undergo some or all of the following procedures for monitoring their health and evaluating their response to treatment:

* Medical history and review of medications
* Physical examination
* Measurement of vital signs (pulse rate, blood pressure, breathing rate and temperature)
* Review of dietary maintenance
* Measurements of height, weight, and waist circumference
* Measurement (with ruler) and photographs of non-Achilles xanthoma
* X-ray of Achilles tendon
* Blood draw and urine collection
* Pregnancy test for women of childbearing potential

DETAILED DESCRIPTION:
Homozygous Sitosterolemia is an inherited, autosomal recessive disorder of sterol metabolism. Patients with homozygous sitosterolemia experience accelerated atherosclerosis with initial coronary heart disease (CHD) events occurring in childhood. Plasma concentrations of sitosterol and other dietary plant sterols are markedly elevated in homozygous sitosterolemic patients, and are characteristic of this disorder. Sitosterolemic individuals demonstrate a range of abnormalities in sterol absorption, metabolism, and excretion. Recent reports have shown that sitosterolemia can result from mutations in 1 of 2 ATP-binding cassette half-transporters (ABCG5 or ABCG8), which are responsible for regulation of non-cholesterol sterols in the body.

Current treatment of homozygous sitosterolemia consists of ezetimibe 10 mg, dietary restriction of plant and shellfish sterols, as well as the use of bile salt binding resins. Ezetimibe is the first member of a new class of cholesterol-lowering agents that inhibits the intestinal absorption of cholesterol and structurally-related noncholesterol sterols (plant sterols) across the intestinal wall. Importantly, ezetimibe is not an inhibitor or inducer of CYP450, reducing the potential for drug-drug interactions which renders ezetimibe a particularly appealing candidate with other drugs. Ezetimibe has proved to be generally safe and well-tolerated as monotherapy or when coadministered with statins, with an overall clinical adverse experience profile similar to placebo. In clinical studies with hypercholesterolemic patients, ezetemibe doses ranging from 0.25 to 40 mg daily for periods of 8 to 12 weeks were more effective than placebo in lowering plasma TC and LDL-C concentrations. There were no dose-related increase in adverse experiences or laboratory abnormalities in these studies. We will investigate whether a higher dose of ezetimibe is safe and efficacious in lowering plant sterols in patients with sitosterolemia.

ELIGIBILITY:
INCLUSION CRITERIA:

To be enrolled into this study, patients must meet all of the following criteria:

1. Patient is at least 18 years of age and no greater than 85 years of age as of Visit 1.
2. Patient has a diagnosis of homozygous sitosterolemia, with a history of a plasma sitosterol concentration greater than 5 mg/dL (0.13 mmol/L).
3. Patient has been on an ongoing stable regimen of ezetimibe 10 mg daily for at least 6 months prior to Visit 1.
4. If patient is currently on a treatment for sitosterolemia (in addition to ezetimibe 10 mg), treatment regimen must be stable for at least 4 weeks prior to visit 1.

   Note: Treatments may include bile salt binding resins, statins, and/or apheresis.
5. Patient must be willing to maintain their current treatment regimen for the duration of the study.
6. Patient must be on a stable diet for at least 4 weeks prior to visit 1.
7. Patient must be willing to maintain this diet for the duration of the study.
8. Patient is a man or postmenopausal woman. Patient is a premenopausal woman who is either surgically sterilized or highly unlikely to conceive, and has a negative urine beta-hCG pregnancy test within 72 hours prior to the start of study treatment.

Note: Highly unlikely to conceive is defined as a woman who: (1) has vasectomized partners, or (2) has a copper intrauterine device (IUD) in place for greater than 3 months without complaint, or (3) abstains from heterosexual intercourse, or (4) agrees to use a double-barrier method of contraception, or (5) is using noncyclical oral contraceptive.

EXCLUSION CRITERIA:

1. Patient has a condition which, in the opinion of the investigator, might pose a risk to the patient, interfere with participation in the study, or does not meet criteria for this protocol.

   MEDICAL HISTORY AND LABORATORY ABNORMALITIES PRIOR TO RANDOMIZATION:
2. Patient has clinically significant laboratory abnormalities at visit 1 and/or last available laboratory results prior to visit 2:

i. ALT (SGPT) greater than or equal to 3 x ULN (75 mU/mL or 75 IU/L).

ii. AST (SGOT) greater than or equal to 3 x ULN (66 mU/mL or 66 IU/L).

iii. TSH greater than 6 microIU/mL or 6mIU/L - or change in medication for hypothyroidism within 6 weeks prior to visit 1.

iv. CPK greater than or equal to 3 x ULN (360 mg/dL or 360 IU/L) and persistent elevation at redraw with muscle symptoms consistent with myopathy.

c. Patient has known hypersensitivity of contraindication to ezetimibe.

d. Patient is breast feeding.

e. Patient's weight is less than 40 kg.

f. Patient has been treated with any other investigational drug within 30 days prior to visit 1.

PROHIBITED MEDICAL CONDITIONS:

g. Patient has uncontrolled cardiac arrhythmias.

h. Patient has had unstable angina pectoris within 1 month of visit 1.

i. Patient has severe/unstable peripheral vascular disease.

j. Patient has had symptomatic carotid disease (transient ischemic attack, stroke) within 1 month of visit 1.

k. Patient had a myocardial infarction within 1 month of visit 1.

l. Patient had a coronary artery bypass surgery, or other invasive coronary procedure within 1 month of visit 1.

m. Patient has a very poorly controlled Type 1 or Type 2 diabetes mellitus (HbA1c at visit 1 greater than 10%), or has had antidiabetic regimen changed within the 8 weeks prior to visit 1.

n. Patient has uncontrolled hypertension (systolic BP greater than 180 mm Hg and/or diastolic BP greater than 110 mm Hg).

o. Patient has impaired renal function (creatinine greater than 2.0 mg/dL or 176.80 micromol/L), or nephritic syndrome at Visit 1.

p. Patient has active or chronic hepatobiliary disease or hepatic disease.

q. Patient is known to be positive for human immunodeficiency (HIV).

r. Patient has a history of severe psychiatric illness, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.

s. Patient had cancer within the past 5 years (except for successfully treated basal and squamous cell carcinomas of the skin).

CONCOMITANT MEDICATIONS/TREATMENTS:

t. Patient is on a statin and is treated with, or likely to require treatment with, an agent that has precautions or contraindications to concomitant use with the statin.

Note: These agents include those with known interactions with statins: antifungal azoles (itraconazole and ketoconazole), macrolide antibiotics (erythromycin and clarithromycin), nefazodone, verapamil, amiodarone, and protease inhibitors.

u. Patient is taking oral corticosteroids UNLESS patient uses as stable replacement therapy for pituitary/adrenal disease. For these indications, patients must be on a stable regimen for at least 3 months prior to visit 1.

v. Patient is on a thiazide diuretic UNLESS treated with a stable regimen for at least 6 weeks prior to visit 1, and expected to remain stable for the duration of the study.

w. Patient had ileal bypass surgery within 3 months prior to visit 1.

x. Patient is currently taking margarines containing phytosterols/phytostanols or other supplements/medications known to increase sitosterol and campesterol concentrations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3
Dates: Start 2004-12; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bhattacharyya AK, Connor WE. Beta-sitosterolemia and xanthomatosis. A newly described lipid storage disease in two sisters. J Clin Invest. 1974 Apr;53(4):1033-43. doi: 10.1172/JCI107640. PMID 4360855
- [Background] Salen G, Shefer S, Nguyen L, Ness GC, Tint GS, Shore V. Sitosterolemia. J Lipid Res. 1992 Jul;33(7):945-55. PMID 1431587
- [Background] Salen G, Horak I, Rothkopf M, Cohen JL, Speck J, Tint GS, Shore V, Dayal B, Chen T, Shefer S. Lethal atherosclerosis associated with abnormal plasma and tissue sterol composition in sitosterolemia with xanthomatosis. J Lipid Res. 1985 Sep;26(9):1126-33. PMID 4067433